CLINICAL TRIAL: NCT03244423
Title: Tranexamic Acid in Cyanotic Heart Defects: a Risk-benefit Analysis.
Brief Title: Tranexamic Acid in Cyanotic Heart Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Profossor of Anesthesiology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB0000879560
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Hemorrhage
Keywords: Pediatric; Cyanotic heart disease; Tranexamic acid; Postoperative blood loss
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): In control group will receive normal saline,
  Interventions: Drug: Normal saline at induction; Drug: Normal saline infusion; Drug: topical normal saline
- Group 2 (Active Comparator): Intravenous Tranexamic acid group will received Intravenous 50 mg / kg followed by infusion of 1 mg/kg/hr for six hours
  Interventions: Drug: Intravenous tranexamic acid; Drug: infusion tranexamic acid; Drug: topical normal saline
- Group 3 (Active Comparator): the topical Tranexamic acid group will receive 50 mg / kg poured before sternal closure.
  Interventions: Drug: Normal saline at induction; Drug: Normal saline infusion; Drug: topical tranexamic acid

INTERVENTIONS:
Drug: Normal saline at induction — 0.5 ml/kg
  Arms: Group 1; Group 3
Drug: Normal saline infusion — 1ml/kg/hr. during surgery for six hours
  Arms: Group 1; Group 3
Drug: Intravenous tranexamic acid — 50 mg/kg
  Arms: Group 2
Drug: infusion tranexamic acid — 1mg/kg/hr infusionfor 6 hours
  Arms: Group 2
Drug: topical tranexamic acid — 50 mg/kg added to the normal saline 2 ml/kg into the pericardial cavity before sternal closure
  Arms: Group 3
Drug: topical normal saline — 2 ml/kg into the pericardial cavity before sternal closure
  Arms: Group 1; Group 2

SUMMARY:
The use of antifibrinolytic agents such as to reduce blood loss in congenital cardiac surgery has been described in many studies

DETAILED DESCRIPTION:
40 patients in each one of the three groups; In control group will receive normal saline, Intravenous Tranexamic acid group received 50 mg / kg intravenousely followed by of 1 mg/kg/hr.for six hours. The topical Tranexamic acid group will have 50 mg / kg of tranexamic poured into the pericoredial cavity. in the first 24 hours we will measure the total blood loss and transfusion requirements. Complate blood picture and coagulation studies will be recorded. the occurrence of re-exploration for excess bleeding, or adverse events.

ELIGIBILITY:
Inclusion Criteria:

2 to 12 years cyanotic cardiac disease with cardio pulmonary bypass

Exclusion Criteria:

Previous cardiac surgery any operation within 48 hr., previous inotropes or mechanical vention aprotinin exposure Liver or renal impairment Coagulation or hemostatic dysfunction within the last 7 days before surgery.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
postoperative blood loss | within the first 24 hours
  Blood loss will be measured within first 24 hr.

SECONDARY OUTCOMES:
total blood transfusion | within the first 24 hours
  ml/kg
the interval from protamine to skin closure | within the first 24 hours
  the interval from protamine to skin closure
the length of ICU stay | within the first month
  by days

CONTACTS AND LOCATIONS:
Overall Officials: Sayed k Abd-Elshafy, MD, Principal Investigator — Associate profossor of anesthesiology
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
UNDECIDED